CLINICAL TRIAL: NCT06701942
Title: Multiple-Family Group Intervention Programming to Improve Mental Health of Adolescents Living With HIV/AIDS in Ghana: An Implementation Science Study Protocol.
Brief Title: Multiple-Family Group Intervention Programming to Improve Mental Health of Adolescents Living With HIV in Ghana: An Implementation Science Approach
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ghana (Other)
Responsible Party: Principal Investigator, Dorothy Serwaa Boakye, Ms, University of Ghana
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: POS-24-07; POS-24-07 (Other Grant/Funding Number: Science for Africa Foundation)
Record Dates: First submitted 2024-11-19; First posted 2024-11-22 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Depressive Disorder; Anxiety Disorder (Panic Disorder or GAD)
Keywords: Multiple family group therapy; Adolescents; HIV/AIDS; Depression; Anxiety
MeSH Terms: conditions — Depressive Disorder; Anxiety Disorders; Panic Disorder; Generalized Anxiety Disorder; Acquired Immunodeficiency Syndrome; Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multiple family group therapy intervention arm (Experimental): ALHIV and their families will be invited to participate in 16 program sessions, each lasting 90 minutes, and will be held on clinic days over a period of 14 weeks.
  The MFG will combine group discussions and activities fostering support, learning and interaction both within the family and among families. The MFG intervention will be delivered by parent peers and community health workers trained by the study team
  Interventions: Other: Multiple family group intervention therapy
- Control Arm (No Intervention): Clinic allocated to the control group will continue with treatment as usual. This group will not receive the MFGT until after the study period when they may be considered to also receive the intervention to ensure all participants eventually benefit from the program. Until then, the control group will receive the usual standard of care including adherence counselling, adherence support, health education and medical care.

INTERVENTIONS:
Other: Multiple family group intervention therapy — Overview The intervention will be implemented at designated clinics where adolescents living with HIV/AIDS (ALHIV) and their families currently receive care. These sites will provide the MFG intervention alongside standard care services. All eligible adolescents and their family members who consent to participate will be included in the intervention group.
  Program Structure The MFG intervention consists of 16 structured sessions, each running for 90 minutes. Sessions will be scheduled to coincide with clinic days over a 14-week period to maximize accessibility and attendance. Parent peers and community health workers, trained by the research team, will facilitate these group sessions.
  Session Format Sessions on the MFGT will begin with introducing participants to one another, the facilitators, and the program curriculum. Subsequent sessions will concentrate on areas such as respectful communication, support, resilience building, problem-solving, conflict resolution, stress management
  Arms: Multiple family group therapy intervention arm

SUMMARY:
When young people living with HIV don't get the mental health support they need, it can lead to a lot of problems. Not only do they suffer from mental health issues, but it also makes it harder for them to stick to their HIV treatment, practice safe sex, go to school regularly, and do well in their studies.

Because of these challenges, experts are urging that we take action to address the mental health needs of these adolescents. They believe that our healthcare system should provide a more comprehensive approach that includes mental health services for these young people. This would not only improve their HIV treatment but also give more people access to mental healthcare around the world.

Being a teenager with HIV is especially difficult, so it's crucial they get the right support, including help with their mental health, to navigate this stage of life. However, many studies show that mental health issues in young people living with HIV, especially in poorer areas, are often ignored. These places often have underfunded and poorly organized healthcare systems, making it even harder to address these problems.

There have been significant advances in treating and preventing HIV, and with the right medication, young people with HIV can now live almost as long as those without the virus. Ghana, like many other countries, has committed to the global goal of ensuring that 95% of people living with HIV are diagnosed, 95% of those diagnosed start treatment, and 95% of those on treatment achieve and maintain low levels of the virus. But these goals are hard to reach without addressing the significant mental health and substance abuse issues faced by adolescents living with HIV.

In Ghana and other low-resource areas, the healthcare system is struggling. Mental health services are rarely included in the basic healthcare that young people living with HIV receive. Most psychiatric units in hospitals are underfunded, so these young people are often referred to specialized hospitals for mental health support. However, financial difficulties, distance, and other barriers prevent many from accessing these services, leaving their mental health needs unmet.

To address this issue, it's essential to integrate mental health services into primary care for adolescents living with HIV. One promising approach is the Multiple Family Group Therapy (MFGT), which could provide much-needed support in these settings.

Multiple Family Group Therapy (MFGT) is a very affordable way to address the emotional and social challenges faced by young people living with HIV and their families. It's a proven method that's listed in the U.S. national registry of effective programs because it uses minimal resources to achieve positive mental health outcomes for many participants.

MFGT was initially designed to help children with behavior problems and their parents, but it has since been used to address a wide range of issues like depression and anxiety in different groups, including people living with HIV. The program is structured and combines group and family therapy, focusing on building skills and improving family dynamics through what are called the 4Rs (Rules, Responsibility, Relationship, and Respectful communication) and 2Ss (Stress and Social support).

The main goal of MFGT is to create a space where families who are dealing with similar challenges can support each other and learn together, all with the aim of improving mental health and behavior. The program helps participants stay engaged with healthcare services, stick to their treatment, reduce symptoms, prevent relapses, and improve their overall quality of life.

Although MFGT was developed in the West and is based on several theories like family systems and social learning, it has been successfully adapted for use in low-resource settings like Ghana. It's particularly appealing in these areas because it can be facilitated by non-professionals such as lay counselors, community health workers, or even parents. This aligns with the World Health Organization's strategy of task-shifting, which involves training non-mental health professionals to provide basic mental health support.

DETAILED DESCRIPTION:
Globally, 38.4 million people are living with HIV, of which 1.7 million are children aged 0-14 years (UNAIDS, 2022). Sub-Saharan Africa contributes substantially to the HIV burden, reflected in the high HIV prevalence, mortality and morbidity (Kharsany & Karim, 2016). Relating to Ghana, about 1.7% of population is living with HIV, with adolescents aged 15-19 years contributing to 0.7% of the HIV burden (Agyemang et al., 2020). The diagnosis of HIV potentiates a cascade of mental health problems that impact all aspect of HIV prevention, treatment/management. This vulnerability is significantly elevated in adolescents who have heightened risk for mental health problems owing to their developmental stage (Wright et al., 2021). In a recent global meta-analytic study, the prevalence of depression among ALHIV was 26.07%, with females (32.15%) and older adolescents aged 15-19 years (37.09%) recording the highest rate than males (25.07%) and younger adolescents aged 10-14 years (29.82%), respectively (Ayano et al., 2021).

Focusing on SSA, a recent systematic review found that 25% ALHIV screened positive for any psychiatric disorder, whereas 30-50% presented with emotional, behavioral difficulties or significant psychological distress (Dessauvagie et al., 2020). Despite the paucity of epidemiological studies in Ghana, existing evidence suggests that ALHIV suffer from discrimination and rejection, ushering them into profound psychological distress such as suicidal thoughts and hopelessness (Doat et al., 2021) that often culminate into poorer psychosocial adjustment (Doku, 2010). Unaddressed mental health problems in ALHIV not only contribute to mental health burden but also negatively impact on treatment adherence, prevention of HIV through adoption of safe sexual practices and behaviors, school attendance and academic achievement (Remien et al., 2019).

In view of the above, analysts have called for a proactive response to the mental health issues in ALHIV(Bhana et al., 2021). In particular, the healthcare systems has been admonished to provide integrated healthcare to ALHIV that includes mental health (Dessauvagie et al., 2020; Vreeman et al., 2017). Doing so would not only strengthen HIV prevention and care outcomes, but it would additionally improve global access to mental healthcare (Remien et al., 2019). Indeed, living with HIV as an adolescent raises the exigency for effective support and guidance, including addressing mental health issues, to ensure they traverse through this developmental stage (Hodgson et al., 2012). However, the literature is replete with the general neglect of mental health problems in ALHIV, particularly in low resource settings where investment in and delivery of mental health are notably poor and disorganized (Essien & Asamoah, 2020). Significant advances have been made in the prevention and treatment of HIV. For example, adolescents diagnosed with HIV can expect a near normal life span given access and adherence to combination anti-retroviral therapy (cART)(Mills et al., 2011; Teeraananchai et al., 2017). Ghana, like other countries have subscribed to the Joint United Nations Programme on HIV/AIDs goal of 95-95-95 call for 95% of people living with HIV (PLWH) to be diagnosed, with 95% of them initiating cART, and 95% of those on cART to achieve and sustain viral suppression through adherence to the treatment. However, these gains will not be achieved without addressing the significant mental and substance use problems among ALHIV(Remien et al., 2019). The lack of research and support for mental health needs in Ghana and other resource-limited settings presents an enormous burden for which cost-effective solutions are urgently needed (Vreeman et al., 2017).

The Multiple Family Group Therapy (MFGT) is an extremely cost-effective interventions that has the tendency to address psychosocial burden holistically among ALHIV and their significant others simultaneously. Listed on the national Registry of evidence-based programs in the US, the MFGT uses relatively minimal resources to achieve positive mental health outcomes for different participants. It was originally developed to target children with disruptive behavior disorders, their parents and service providers but has since been applied to address a range of psychopathological behaviors such as depression, anxiety in different population, including individuals living with HIV(Sensoy Bahar et al., 2020). As a structured program and a hybrid of group and family interventions, the MFGT is focused on improving skills and family processes referred to as 4Rs (Rules, Responsibility, Relationship and Respectful communication) and 2Ss (Stress and Social support). The key therapeutic aim of MFGT is to foster mutual support and learning between families who face similar difficulties and are united by a common goal of improving mental health and behavioral outcomes (Loh et al., 2021). It aims to support engagement with healthcare service, treatment adherence, symptoms reduction, relapse prevention, and quality of life. The MFGT is a Western-based model with strong theoretical underpinning, been a derivative of multiple theories such as family systems, structural family, and social learning theories. It is also anchored in psychoeducation and social group work. The MFGT is attractive in low resource settings such as Ghana given that it has been successfully facilitated by lay counsellors, community health workers, village health team and/or parent peers(McKay et al., 2004; Mellins et al., 2014). This is consistent with the task shifting strategy proposed by the WHO to address mental health problems by empowering non-mental health professionals to provide essential and basic mental health support(Adjorlolo et al., 2019).

The major caveats in relation to the application of the MFGT in Ghana are two-fold. First, the MFGT is formulated based on predominantly individualistic, western family principles, processes and practices that starkly contrast family systems in predominantly collective societies, including Ghana. This questions the application of the MFGT in Ghana without recourse to Ghanaian family systems and practices(Asampong et al., 2021; Sensoy Bahar et al., 2020); an observation that necessitates the adaption of the MFGT to increase its sensitivity to the local settings and family systems in Ghana. Although some versions of the MFGT have been incorporated into a family-based HIV prevention intervention (i.e., CHAMP program) in South Africa (McKay et al., 2004; Mellins et al., 2014) and family focused economic strengthening intervention (SUUBI program) in Uganda(Ssewamala et al., 2014), this is the first attempt to wholly adapt the MFGT to address mental health and psychosocial issues in ALHIV in SSA, focusing on Ghana. Previous effort to adapt the MFGT in Uganda has centered on adolescents with disruptive behaviors disorders in educational settings; a population that is functionally and psychological distinct from ALHIV, including family structures and functioning. Besides, none of the previous efforts were aimed at healthcare system strengthening to deliver integrated health services that include mental health support. Owing to the limited human resource, finance and logistics, the healthcare system in Ghana, just like other countries in SSA, is fragmented mostly at the primary level. Mental health services are barely integrated into the primary healthcare for ALHIV. Most of the psychiatric units of the Ghanaian hospitals are poorly resourced, making referrals of ALHIV in need of mental support to psychiatric hospitals the most viable option. However, financial problems and geographic barriers and others limit the utilization of the referral system, leaving the mental health of ALHIV unaddressed. This demands the integration of mental health support system into the primary care for ALHIV; the MFGT holds significant prospects in this regard.

This study aims to adapt, implement, and evaluate the effectiveness of the MFG intervention to improve mental health outcomes among adolescents living with HIV in Ghana using an implementation science approach. The specific objectives of the study are:

To culturally adapt an existing MFG intervention for use with HIV-positive adolescents and their families in Lower Manya Krobo, addressing mental health outcomes and treatment adherence.

To implement the adapted MFG intervention in selected healthcare facilities in Lower Manya Krobo.

To evaluate the effectiveness of the adapted MFG intervention in improving mental health outcomes, and enhancing treatment adherence The study will be carried out in the Atua and Asesewa communities within the Lower Manya-Krobo district. This district is chosen due to its high HIV prevalence (5.6% compared to the regional prevalence of 2.8%) and the presence of established HIV care facilities.

The entire study will be carried out in three phases. Phase one is the Adaptation phase which will involve Cultural adaptation of the MFG intervention through stakeholder engagement and focus group discussions. Phase two is the Pilot implementation phase which will involve the implementation of the adapted intervention in selected healthcare facilities. Phase three is the evaluation phase which will involve the process, impact and outcome assessment of intervention effectiveness.

The Theory of Triadic Influence (Bell et al., 2002) will guide the cultural and contextual adaptation process. This theory argues that childhood behavioral challenges are products of multiple streams of influence thus the intrapersonal stream linked to qualities inherent in the adolescent, the social normative stream linked to the immediate family context and the adolescent, and cultural attitudinal stream linked to the sociocultural environment (Flay & Petraitis, 1994). We will supplement the Theory of Triadic Influence with frameworks taken from Social Action Theory (Ewart, 1991), which is a model of behavior change. The adaptation coding framework by Stirman et al., (2013), will be used to document the modifications made to the 4Rs and 2Ss for the Ghanaian context.

The adaptation process will involve a four-phase stakeholder engagement and collaborative meetings, guided by previous adaption efforts (Asampong et al., 2021; Mellins et al., 2014; Sensoy Bahar et al., 2020) and theories of adaption(Bell et al., 2002; Ewart, 1991; Stirman et al., 2013). Phase 1 is mapping and recruitment of at least 30 stakeholders and initial meetings with stakeholders to create awareness about the project, solicit their views on the scope and expectations of the project and empower them as agents of change to facilitate sustainable collaborations and scale-up of the intervention. Therefore, the powers and influence of each stakeholder is critical to the project. The stakeholders will comprise parents, older family members (e.g., Nephew, Cousin), children/adolescents, family heads, local chiefs and queen mothers, health professionals, including community health officers. The MFGT, focusing on 4Rs and 2Ss, would be presented to the stakeholders to discuss their relevance and application in Ghanaian families. Phase 2 involves a review of the MFGT curriculum/manual. Prior to this, the PI and the research team, with the support of supervisors and other local experts will review the MFGT manual to understand the relevance of its concepts and content for the Ghanaian context. The team will also brainstorm about context-specific activities and examples to be adapted or added. During the review, the stakeholders will be encouraged to note the aspect of the MFGT they have issues with and how the issues can be addressed. These will be discussed with all stakeholders present to arrive at a solution. The stakeholders will address questions such as the number of families for the MFGT, family composition, the timing of intervention delivery, duration and number of sessions, and their opinions about who should lead intervention delivery (i.e., health professionals versus parent peers), location of intervention delivery, the target behaviors for intervention and expected outcome and assessment of outcome. Phase 3 is revision of the MFGT curriculum content based on the inputs, suggestions, and feedback from the stakeholders in phase 2. This is the responsibility of the PI and research team, with the support of project supervisors. Phase 4 is finalization and approval of adapted curriculum/manual. The stakeholders would be invited to review the revised curriculum, ensuring that the content captures all discussions and issues raised in phase 2. Request for new revisions would be tolerated if majority of the stakeholders endorse the revision. This iterative process would be followed until the stakeholders accept the adapted curriculum as reflective of and sensitive to Ghanaian culture and family value systems.

The intervention will be piloted using a pretest-posttest control group design. Two MFGs would be constituted, matched on demographics. They would be randomized into control and intervention groups. The control group will receive the usual care whereas the intervention group will be administered the MFGT. The two MFGs would be selected from facilities or locations that are geographically far apart to guard against contamination of treatment, defined as when participants in another study arm request for all or some of the services in other arms such that the groups are now receiving the same or almost the same interventions. The delivery of the intervention would be underpinned by the adapted MFGT manual/curriculum. The sample size is determined based on the practical difference in expected mean (that is, pre- post-intervention outcome) in the intervention arm. Using the G*power2 computer program (Faul et al., 2007), a significance level (α) of 0.05, power of 80% (β = 0.2), and an allocation ratio of 1:1 for two independent arms of the study, a total of 72 ALHIV is needed to detect an effect of 0.6 (approximately 36 per study arm). We anticipate an attrition/non-response rate of 10% for each arm of the study (i.e., 10% of 36 = approximately 4 additional participants for each study arm). Therefore, a minimum of 80 ALHIV and their families would be recruited for the study, with each study arm requiring a minimum of 40 participants. Previous studies that adopted versions of the MFGT in South Africa included 12 to 20 families (Mellins et al., 2014). Therefore, barring no change in the number of families for a MGFT in the Ghanaian context, a minimum of four MFGs and a maximum of two MFGs for each study arm would be needed to achieve a sample size of 80. Study Outcomes: The main study outcome variable is improvement in mental health and wellbeing, focusing on depressive and anxiety symptoms. Depression and anxiety symptoms would be assessed using the Patient Health Questionnaire (Kroenke et al., 2001) and Generalized Anxiety Disorder (Spitzer et al., 2006), both of which have been validated in Ghanaian adolescents (Adjorlolo, 2019; Anum et al., 2019). The secondary outcome variable is adherence to antiretroviral therapy and it would be measured using the Three-Item Self-Report Measure for Medication Adherence (Wilson et al., 2016). This is crucial as it will establish a connection between mental health and HIV outcomes, highlighting the necessity of implementing mental health interventions.

The last phase of the study which is the evaluation phase will be iterative and formative (Longworth et al., 2024). Attention will be paid to both effectiveness and participants' experiences (Longworth et al., 2023). This phase of the study will be achieved in three steps.

Step 1: Process Evaluation.The primary purpose is to provide information about program improvements; by establishing whether the implementation is proceeding as planned, ie. (Issel, 2004; Hawe, Degeling & Hall, 2003) is the program reaching all members of the target group, are all the materials and components of the program of good quality, are all the planned activities of the program being implemented, are all the participants satisfied with the program. This step will be achieved through questionnaires administration for participants and facilitators. We will also conduct focus group discussions involving participants and facilitators.

Step 2: Impact Evaluation. The primary purpose is to provide information about program improvements; by establishing whether the implementation is proceeding as planned, ie. (Issel, 2004; Hawe, Degeling & Hall, 2003) is the program reaching all members of the target group, are all the materials and components of the program of good quality, are all the planned activities of the program being implemented, are all the participants satisfied with the program

Methods to achieve step 2:

Questionnaires for participants and facilitators Focus groups involving participants and facilitators Checklists and/ or Observations. Step 3: Outcome Evaluation. This measures the long-term effects of the program, i.e., whether it meets its goals; by determining what changes, if any, have occurred in health status and quality of life (Hawe, Degeling & Hall, 2003).

This will be done 3 and 6 months post-intervention Methods to achieve step 3: post-intervention questionnaire for participants. Timing of Assessment: Baseline: Before the intervention begins, Mid-intervention: Halfway through the intervention period, Post-intervention: Immediately after the intervention ends and Follow-up: 3 and 6 months after the intervention

Data analysis: : Independent t-test would be used to assess differences between the arms on mental health outcomes, whereas within group differences (pre-posttest scores) would be investigated using repeated measure analysis. Descriptive statistics would be used to summarize participants demographic and responses to categorical study variables. Chi-square and Pearson correlation would be used to determine the relationship between the study variables. Mediation Analysis using structural equation modelling will be done to account for potential mediators such as family functioning, and stigma.

The data collected from in-depth interviews and focus group discussions would be subjected to a rigorous thematic analytical process guided by Braun and Clarke's (2022) recommendation.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents:

Aged 10-19 years (as per WHO definition of adolescence) Confirmed HIV-positive status Currently receiving antiretroviral therapy (ART) Aware of their HIV status Residing in Lower Manya Krobo district Able to communicate in either English or the local language Willing to participate in group sessions

Caregivers/family:

Primary caregiver of an eligible adolescent participant Aged 18 years or older Aware of the adolescent's HIV status Residing in Lower Manya Krobo district Able to communicate in either English or the local language Willing to participate in group sessions

Exclusion Criteria:

* Adolescents:

Presence of severe cognitive impairment that would prevent participation in group activities Acute psychiatric conditions requiring immediate intensive treatment Current participation in another mental health intervention study Unable to provide assent or obtain caregiver consent

Primary Caregivers/Family:

Presence of severe cognitive impairment that would prevent participation in group activities Acute psychiatric conditions requiring immediate intensive treatment Unable to provide informed consent

Both Adolescents and Caregivers:

Planning to relocate outside of Lower Manya Krobo district within the next 12 months Unable to commit to attending the majority of planned group sessions

Ages: 10 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-01-15 (Estimated); Primary Completion 2025-08-20 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Depression. | Baseline, immediate post intervention and 3, and 6 months follow-up
  Depression will be assessed with the Patient Health Questionnaire-9 (PHQ-9) (Kroenke et al., 2001) which has been validated for use with adolescents and in Ghanaian settings (Adjorlolo, 2019) The PHQ-9 has 9 items, each scored 0-3, with a total score range 0-27 Scores ≥10 indicate moderate to severe depressive symptoms
Anxiety | Baseline, immediate post intervention and 3, and 6 months follow-up
  Anxiety will be assessed with the Generalized Anxiety Disorder-7 (GAD-7) (Spitzer et al., 2006), whic has also been validated for use in Ghanaian adolescents (Anum et al., 2019). The GAD-7 has 7 items, each scored 0-3, with a total score range of 0-21. Scores ≥10 indicate moderate to severe anxiety symptoms

SECONDARY OUTCOMES:
Adherence to Antiretroviral therapy | Baseline, immediate post intervention and 3, and 6 months follow-up
  Adherence will be assessed by the Wilson's 3- item Self-reported adherence measure (Wilson et al., 2016). Participants level of adherence will be marked on a line from 0-100% on a 0-100 scale with zero being the worst adherence, and 100 the best (Wilson et al., 2016)

IPD SHARING:
Plan to Share IPD: Yes
Study description, protocol summary, Arms and interventions, Outcome measures and eligibility.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: The de-identified Individual Participant Data (IPD) and supporting documentation will be made available starting [insert start date, e.g., six months after primary study results are published]. This timeframe ensures adequate time for the study team to finalize and publish the primary findings.
  Data will remain accessible for 5 years after the start date, during which researchers can request access in line with the data-sharing policy. This period may be extended upon review and at the discretion of the study team
Access Criteria: Individual Participant Data (IPD) Access Statement
  Access to Individual Participant Data (IPD) and supporting documentation from this study will be available to qualified researchers for non-commercial, academic purposes that align with the goals of advancing public health and scientific knowledge. The following details describe the access framework:
  Who will be able to access the data? Data access will be granted to researchers affiliated with recognized institutions, universities, or organizations that submit a formal request and demonstrate the scientific merit of their proposed analysis. Applicants must also provide proof of ethical clearance for their secondary analysis and agree to abide by data protection regulations.
  What will they be able to access? Approved researchers will have access to de-identified participant-level data (IPD), which will include demographic, intervention, and outcome variables relevant to the study objectives.

REFERENCES:
- [Derived] Boakye DS, Adjorlolo S. Stakeholder perspectives on contextual barriers to the successful implementation of multiple family group therapy in the Lower Manya Krobo District, Ghana: a qualitative study. BMJ Open. 2025 Sep 8;15(9):e105448. doi: 10.1136/bmjopen-2025-105448. PMID 40921643
- [Derived] Boakye DS, Adjorlolo S. Multiple-family group intervention programming to improve mental health of adolescents living with HIV/AIDS in Ghana: An implementation science study protocol. PLoS One. 2025 Jun 12;20(6):e0325854. doi: 10.1371/journal.pone.0325854. eCollection 2025. PMID 40504853